CLINICAL TRIAL: NCT05515666
Title: The Value of Wearable Electrocardiogram in the Diagnosis of Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020-ZX68
Record Dates: First submitted 2022-06-24; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Electrocardiogram
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Wearable electrocardiogram — All participants will have their ECG monitored at home using a wearable ECG, and then be hospitalized for coronary angiography and quantitative flow fraction to confirm the presence of coronary artery disease.

SUMMARY:
ECG is one of the classic tests for coronary artery disease, but patients with coronary artery disease often have no onset of typical symptoms at the time of consultation, so it is difficult to capture ischemic changes on a conventional ECG. In this study, a diagnostic test was performed to assess the diagnostic value of wearable ECG for coronary artery disease, with the gold standard of coronary angiography and quantitative flow fraction. In addition, we followed up with the enrolled participants for 1 year to assess the relationship between wearable ECG and long-term prognosis.

DETAILED DESCRIPTION:
Background: Patients with suspected coronary artery disease usually have symptoms such as angina, shortness of breath, and fatigue during daily life. But they may have no typical symptom when they arrived at the hospital. If routine examinations and laboratory tests such as electrocardiogram and cardiac markers cannot support the diagnosis of coronary heart disease, patients often need coronary computed tomography angiography or hospitalization for coronary angiography. This advanced diagnostic imaging has several shortcomings such as radiation exposure, long time for the appointment, certain requirements for patient's physical condition (such as exercise ability, good liver and kidney function, etc.), corresponding mental stress and economic burden to the patient. Therefore, for patients with suspected coronary artery disease but cannot be diagnosed by routine examinations, new diagnostic methods that are both safe, accurate, and economical are needed.

Aims: This project intends to assess the diagnostic value of wearable electrocardiograms for coronary artery disease. Patients will take the device home and actively record the electrocardiogram at symptoms onset. The data will be uploaded to the diagnostic center and read by professional cardiologists. The results will be compared with coronary angiography to test its diagnostic efficacy. It is hoped that the diagnosis efficiency of coronary artery disease and patients' experience can be improved.

Operating Procedures:

1. Baseline information was collected from subjects who met the inclusion criteria, including demographic information such as gender and age, chief complaints and past history, outpatient blood pressure values, 12-lead ECG results, baseline results of the wearable ECG, and hematological test results such as myocardial enzyme profile tests. The technician conducts patient education to ensure that subjects are clear about the requirements for use of the wearable ECG and how to upload it, know the process of home monitoring, and reserve contact information for both doctors and patients.
2. Participants lived a normal life at home and used the wearable ECG to collect an ECG once a day in the early morning. If symptoms related to coronary artery diseases, such as chest tightness and chest pain, occur at home, the ECG is recorded immediately using the wearable ECG, and a simple complaint of the attack is selected on the corresponding mobile app and uploaded to the cloud data center. The ECG can be collected and uploaded several times during the onset of symptoms without removing the wearable ECG, and then again after the symptoms have disappeared. If the subject's symptoms do not subside or even worsen during the period, or if the subject feels that he/she needs medical attention, he/she should go to our center or to the nearest hospital for medical treatment in a timely manner. The uploaded ECG will be interpreted by the ECG physician at the diagnostic center for abnormalities.
3. Diagnostic criteria of wearable ECG for myocardial ischemia.

   ① ST-segment depression of horizontal or inferior type ≥ 0.1 mV (1.0 mm), lasting ≥ 1.0 min, with an interval of ≥ 5.0 min between episodes. a significant increase/slowing of the mean heart rate during the episode compared to 10-30 min before the episode (20 beats/min increase or 10 beats/min decrease is recommended as the diagnostic reference cut point), or the concomitant presence ② ST-segment elevation showing ischemic J waves with duration ≥ 1.0 min and the interval between episodes ≥ 5.0 min. The mean heart rate during the episode is significantly increased/decreased compared with 10-30 min before the episode (an increase of 20 beats/min or a decrease of 10 beats/min is recommended as the diagnostic reference cut point) or accompanied by arrhythmias.

   ③ Ischemic evolution of the ST-T on a transient or intermittent basis in the monitoring of the ECG is clinically significant.
4. When the participants were admitted to the hospital, the preoperative examination was first completed to clarify that there were no contraindications to coronary intervention, then coronary angiography was performed and quantitative flow fraction (QFR) was measured, and the need for revascularization treatment was judged by the operator during the intervention. The criteria for the diagnosis of coronary artery disease are QFR ≤ 0.8 in at least one coronary stenosis lesion, or decreased blood flow in the lesion with stenosis ≥ 90% of the vessel diameter. Subjects without meaningful stenosis on coronary angiography were required to undergo loading myocardial perfusion imaging to evaluate microvascular lesions.
5. Follow-up: The end of follow-up is 1 year after hospital discharge. During this period, four follow-up visits were conducted by telephone or outpatient at 30 days, 3 months, 6 months, and 12 months after the subjects were discharged from the hospital. The follow-up visits included major cardiovascular adverse events (all-cause death, total myocardial infarction, stroke, target vessel revascularization, etc.), rehospitalization, and cardiac-related diseases and treatment.

Statistics: The diagnostic results of the wearable ECG were compared with those of QFR, and sensitivity, specificity, positive predictive value, negative predictive value, positive likelihood ratio and negative likelihood ratio, compliance rate, and 95% confidence interval corresponding to each index were calculated. The significance level of the statistical test was taken as 5% bilaterally.

ELIGIBILITY:
Inclusion Criteria:

1. age >=18 years & age <=75 years;
2. with suspected coronary artery disease;
3. with any clinical indication for percutaneous coronary intervention;
4. left ventricular ejection fraction >40%.

Exclusion Criteria:

1. acute myocardial infarction;
2. rheumatic heart disease, malignant arrhythmia;
3. valvular heart disease;
4. thoracic deformities, infections, skin ulcers, allergies, etc. who cannot use wearable ECG;
5. severe hepatic impairment;
6. renal failure;
7. iodine allergy;
8. known pregnancy；
9. inability to provide informed consent；
10. currently participating in another trial before reaching primary endpoint.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected coronary artery disease and cannot get a diagnosis by routine examination such as traditional ECG.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The Diagnostic Yield of wearable electrocardiogram for the diagnosis of obstructive CAD in whole population and in the subgroups including patients of different genders and age groups | an average of 2 year
  The results of wearable electrocardiogram (for example, ST segment change) will be compared with coronary angiography, The diagnostic standard of coronary angiography for obstructive CAD is anatomic coronary narrowing >= 90% or Quantitative Flow Ratio <=80%.

CONTACTS AND LOCATIONS:
Overall Officials: Hongjian Wang, Doctor, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Hongjian Wang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No